CLINICAL TRIAL: NCT04992130
Title: Sport-Related Concussion and Traumatic Lower Body Injury Performance-Based Prevention Program
Brief Title: Sport Concussion Performance-Based Prevention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Brian Benson, Assistant Research Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB21-1027
Record Dates: First submitted 2021-07-20; First posted 2021-08-05 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Concussion, Brain; Traumatic Injury
MeSH Terms: conditions — Brain Concussion; Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention cohort (Experimental): Pre-season supplementary neurologic training program
  Interventions: Behavioral: Pre-season supplementary neurologic training program
- Control cohort (No Intervention): Usual pre-season training program

INTERVENTIONS:
Behavioral: Pre-season supplementary neurologic training program — A two-month standardized, pre-season, supplementary multi-modal training program will be prescribed to 200 athletes (intervention cohort) by a team of experienced sport science and medicine professionals targeting the specific intrinsic risk factors of interest identified in the current concussion and ACL prevention literature.
  Arms: Intervention cohort

SUMMARY:
Sport-related concussions and traumatic lower body injuries (e.g., anterior cruciate ligament (ACL) tears) occur frequently in high-speed and contact/collision sports contributing to significant time loss from training/competition and potentially devastating long-term performance and health consequences. Neurological impairment following a concussive injury may be subtle, but if missed, may have grave consequences in a high-risk, high-speed sporting context. Recent evidence suggests that the risk of lower body musculoskeletal injury is significantly higher for athletes sustaining a sport-related concussion in the three-month to two-year period following injury. Most injury prevention research to date has focused on modifiable extrinsic risk factors; there is a void or gap on modifiable intrinsic risk factors.

The purpose of this study is to:

1. determine the effect of a standardized supplementary pre-season multi-modal neurologic training program, versus usual training, on concussion and/or traumatic lower body injury risk among high-speed/contact/collision sport athletes (primary prevention).
2. determine the effect of a standardized supplementary pre-season multi-modal neurologic training program, versus usual training, on concussion and/or traumatic lower body injury severity (time loss from training/competition measured in days, determined from the date of injury to the date a sport medicine physician medically clears the athlete to return to unrestricted training/competition) (secondary prevention).
3. determine the effect of a standardized supplementary pre-season multi-modal neurologic training program, versus usual training, on neurologic performance.

The investigators hypothesize that athletes completing the standardized supplementary pre-season multi-modal neurologic training program, compared with usual training, will significantly reduce the participants risk and severity of concussion and/or traumatic lower body injury, and significantly improve neurologic performance.

DETAILED DESCRIPTION:
This study will measure multiple neurological systems and brain processes on 400 Canadian high-performance snow sport athletes and elite community ice hockey players in the participants healthy (uninjured) state using reliable assessment technology and techniques. A two-month standardized, pre-season, supplementary multi-modal training program will be prescribed to 200 athletes (intervention cohort) by a team of experienced sport science and medicine professionals targeting the specific intrinsic risk factors of interest identified in the current concussion and ACL prevention literature. The control cohort of 200 athletes will carry out their usual pre-season training programs. At the completion of the two-month training period, the standardized neurological outcome measures completed at baseline will be repeated on all athletes.

ELIGIBILITY:
Inclusion Criteria:

1. participation at the Canadian Senior National, National Development, Provincial, Sport School, Academy or Club levels of competition for skiing and snowboarding athletes, or participation in the Canadian Sport School Hockey League or Hockey Calgary U16 or first year U18 ice hockey levels of competition for hockey players between August 2021 and April 2023;
2. male or female;
3. assessed for a concussion or traumatic lower body injury that was sustained during an organized training session/practice or competition/game and diagnosis confirmed by a sport medicine physician; and
4. written informed consent to participate during the 2021-2022 and 2022-2023 seasons.

Exclusion Criteria:

1. previous history of neurological issues such as stroke, seizure, and/or congenital intracranial abnormalities, or non-fully resolved concussion or traumatic lower body injury sustained in the 3-month period prior to the initiation of study; and
2. non-sport-related concussions or traumatic lower body injuries.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of sport-related concussion injuries sustained by participants during the study period as diagnosed by the study physician. | Two years
  Sport-related concussion diagnosis will be based on clinical judgment by an experienced sport medicine physician based on participant self-report of post-traumatic clinical signs and symptoms, comprehensive neurological examination, and the Sport Concussion Assessment Tool (SCAT5).
Number of acute traumatic lower body injuries sustained by participants during the study period as diagnosed by the study physician. | Two years
  Acute, traumatic lower body injury to the hip, thigh, knee, leg, ankle, foot including, but not limited to, fracture including avulsion fracture, labral tear, muscle contusion/tear, tendon strain/tear, ligament sprain/tear, meniscus tear, subluxation/dislocation, chondral injury or nerve injury diagnosed by study physician.

SECONDARY OUTCOMES:
Sensorimotor function as measured by the Kinesiological Instrument for Normal and Altered Reaching Movements (Kinarm, Kingston, Ontario, Canada) end-point robotic standard tasks. | Mean change from baseline sensorimotor function on the Kinarm Standard Tasks at 8-weeks post pre-season training.
  Kinarm Standard Tasks:
  1) Visually Guided Reaching task examines visuomotor capability through parameters such as reaction time, movement speed, movement direction and smoothness.
  2. Position Matching task examines proprioception through parameters such as absolute matching error and variability.
  3. Object Hit task examines bimanual motor ability and visuospatial attention through parameters such as total hits, workspace use of each hand and movement speed.
  4. Object Hit and Avoid task examines attention, rapid motor selection and inhibition through parameters such as distractor hits, workspace use of each hand and movement speed.
  5. Trail Making B task examines attention and task-switching through parameters such as total test time and number of errors.
Neuromuscular function as measured by force plates and motion sensor. | Mean change from baseline neuromuscular function on the neuromuscular tasks and wearable sensor at 8-weeks post pre-season training.
  Neuromuscular Assessments:
  1) between-limb vertical jump force-time asymmetry testing, 2 hamstring/quadriceps rapid force production and maximal strength testing, 3) lower body power endurance, workload capacity and fatigue tolerance, 4) hip muscle strength and landing abilities, 5) quadriceps and hamstring rate of force development in the vertical countermovement jump, 6) clinical grade wearable sensor (PROTXX) attached to the participant's mastoid using a disposable medical adhesive directly measuring linear and rotational accelerations of the body.
Visual function as measured by the RightEye eye-tracking system. | Mean change from baseline visual function on the RightEye eye-tracking tasks at 8-weeks post pre-season training.
  RightEye is a Food and Drug Administration (FDA) approved healthcare technology designed to assess vision and associated brain health (i.e., fixation, eye teaming, object tracking, eye-hand coordination, reaction time).
Cognitive function as measured by the computer-based Immediate Post-Concussion Assessment and Cognitive Test (ImPACT). | Mean change from baseline cognitive function on the ImPACT neuropsychological composite scores at 8-weeks post pre-season training.
  Measurement of memory, attention span, visual and verbal problem solving function using four composite scores (Verbal Memory Composite, Visual Memory Composite, Visual Motor Speed Composite, and Reaction Time)
Dynamic neck strength as measured by the TopSpin360 neuromuscular neck-strengthening device. | Mean change from baseline dynamic neck strength at 8-weeks post pre-season training.
  The TopSpin360 device has an electronic counter that counts the number of revolutions and calculates the speed of the weight in revolutions per minute (RPM).

CONTACTS AND LOCATIONS:
Locations (1):
- Benson Concussion Institute, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No